CLINICAL TRIAL: NCT01469143
Title: A Trial Investigating the Pharmacokinetic Properties of Formulations of NN1218 in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1218-3977; 2011-004081-15 (EudraCT Number); U1111-1123-6692 (Other: WHO)
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NN1218 (Experimental)
  Interventions: Drug: Faster-acting insulin aspart
- insulin aspart (Active Comparator)
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: Faster-acting insulin aspart — Each subject will randomly be allocated to a treatment sequence consisting of 9 dosing visits during which the subject will receive 8 single doses of different formulations. For all investigational medicinal products the dose levels will be 0.2 U/kg body weight (BW). The trial products will be administered subcutaneously (under the skin).
  Other Names: NN1218
  Arms: NN1218
Drug: insulin aspart — At one of the scheduled visits, the subject will receive a single dose of insulin aspart. The dose level will be 0.2 U/kg body weight (BW). The trial products will be administered subcutaneously (under the skin).
  Arms: insulin aspart

SUMMARY:
This trial is conducted in Europe. The purpose of this trial is to compare the pharmacokinetic properties (the exposure of the trial drug in the body) of different formulations of NN1218.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus for more than 12 months
* Treated with multiple daily insulin injections or continuous subcutaneous insulin infusion (CSII) for more than 12 months
* Body mass index (BMI) between 18.0-28.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Subjects who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to trial start
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day)
* Not able or willing to refrain from smoking and use of nicotine gum or transdermal nicotine patches during the inpatient period

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Area under the serum insulin aspart concentration-time curve | From 0 to 1 hour

SECONDARY OUTCOMES:
Area under the serum insulin aspart concentration-time curve | From 0 to 12 hours
Maximum observed serum insulin aspart concentration | From 0 to 12 hours
Time to maximum observed serum insulin aspart concentration | From 0 to 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com